CLINICAL TRIAL: NCT04886271
Title: A Multicenter Phase II Clinical Study of Recombinant Humanized Anti-CD47 / PD-1 Bifunctional Antibody HX009 Injection in the Treatment of Advanced Solid Tumors
Brief Title: Recombinant Humanized Anti-CD47 / PD-1 Bifunctional Antibody HX009 Injection in the Treatment of Advanced Solid Tumors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Waterstone Hanxbio Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HX009-II-01
Record Dates: First submitted 2021-05-05; First posted 2021-05-14 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HX009 (Experimental)
  Interventions: Drug: HX009

INTERVENTIONS:
Drug: HX009 — Eligible participants will receive HX009 treatment at 5mg/Kg via IV infusion over 60-120 minutes, and the scheduled dosing cycle is once every 2 weeks.

SUMMARY:
This is a multi-center phase II clinical trial to evaluate the anti-tumor activity and safety of HX009 in subjects with advanced solid tumors.

DETAILED DESCRIPTION:
The present study is comprised of two parts: the efficacy estimation part and the key phase II part. In the first part, subjects with unresectable locally advanced or metastatic solid tumors (confirmed by histology or pathology) will be enrolled. Tumor types of special interest include biliary cancers, head and neck cancers, esophageal cancers, sarcoma, and malignant mesothelioma, and at least 8 subjects will be enrolled for each of these tumor types. Subjects with biliary cancers and other tumor types based on the efficacy data of the first part will be enrolled in the second part of the study.

Subjects will receive HX009 via intravenous infusion at 5 mg/Kg once every 2 weeks. Treatment will continue until loss of clinical benefit at the discretion of the investigator, or intolerable toxicity, or withdrawal of consent, or disease progression, or death, or loss of follow-up (whichever occurs first). The maximum duration of treatment with HX009 is one year.

Tumor evaluation is conducted by the investigator according to the Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) and immune RECIST (iRECIST), and is repeated every 6 weeks. Adverse events (AEs) are graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18 to 75 years, inclusive;
2. Eastern Cooperative Oncology Group performance status of 0 to 1;
3. Having unresectable locally advanced or metastatic solid tumor (confirmed by histology and cytology);
4. Participants must have failed the standard treatment (due to either disease progression or intolerable toxicity) or the standard of care had not been established for the specific condition;
5. Measurable extracranial lesion based on Response Evaluation Criteria In Solid Tumors (RECIST) 1.1;
6. Life expectancy ≥12 weeks;
7. For prior anti-tumor therapies, the following conditions must be met:

   * The interval between local radiotherapy or radiotherapy for bone metastasis and the first dose is ≥2 weeks;
   * The interval between the last dose of previous chemotherapy, immunotherapy (including PD-1, PD-L1 or CTLA-4 antibodies), biological therapy (tumor vaccines, cytokines, or anti-cancer growth factors) and the first dose of HX009 is ≥4 weeks (The interval between the last dose of small molecule targeted drugs and the first dose of HX009 is ≥2 weeks);
   * The interval between the last dose of anti-cancer Traditional Chinese Medicine and the first dose of HX009 is ≥ 2 weeks;
   * Has had previously serious adverse reactions (pneumonia or myocarditis) related to previous PD1/PDL1or CTLA-4 inhibitors that preclude their treatment according to the investigator's criteria;mmune-related adverse reactions must be restored to Grade 1 except for adverse endocrine system reactions;
8. Participants with asymptomatic central nervous system (CNS) metastases are eligible only if they have no evidence of progression by imaging for at least 12 weeks prior to the first dose of HX009 and are not using corticosteroids;
9. Appropriate organ functions according to the following laboratory tests :

   * Absolute neutrophil count (ANC)≥1.5 × 10^9/L
   * Absolute white blood cell count (WBC) ≥3.0×10^9/L
   * Platelet count ≥90 × 10^9/L
   * Hemoglobin ≥90 g/L
   * Serum creatinine≤1.5 upper limit of normal (ULN)
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 × ULN , ALT and AST ≤5 × ULN for subjects with liver metastases or liver cancer
   * Serum Total bilirubin (TBIL) ≤1.5 × upper limit of normal (ULN)
   * International normalized ratio (INR) ≤ 2 x ULN, or activated partial thromboplastin time (APTT) ≤ 1.5 x ULN (except for patients receiving anticoagulant therapy) ;
10. Reproductive males or females who are likely to become pregnant must use highly effective contraceptive methods (such as oral contraceptives, intrauterine contraceptives, sexual control or barrier contraceptives combined with spermicides) during the trial, and continue contraception for 6 months after the last dose of HX009;
11. Participants must be willing and able to provide written informed consent for the study, and have good compliance;

Exclusion Criteria:

1. Participants having a known additional malignancy within 5 years before enrollment, except for malignancies with low risk of metastasis and death (5-year survival rate> 90%), such as completely resected basal cell or squamous cell skin cancer, or cervical carcinoma in situ, or superficial bladder cancer,early breast cancer with low risk of recurrence, etc;
2. Adverse reactions related to previous treatment that failed to recover to CTCAE 5.0 ≤ grade 1 (chemotherapy-induced alopecia or grade 2-3 peripheral neurotoxicity are eligible; immune-related grade 2-3 hypothyroidism is eligible)；
3. Participants with active or history of autoimmune diseases are ineligible, except for the following conditions:

   * Participants with type 1 diabetes who are in stable condition after using a fixed dose of insulin;
   * Autoimmune hypothyroidism requiring only hormone replacement therapy;
   * Autoimmune skin diseases that do not require systemic treatment (such as eczema, skin rashes that account for less than 10% of the body surface, or psoriasis without ophthalmological symptoms);
4. Participants expected to undergo major surgery within 28 days before the planned first dose of HX009;
5. Participants receiving systemic corticosteroids equivalent to >10 mg prednisone/day or other immunosuppressive drugs within 14 days before the first administration of HX009, except for the following conditions:

   * Participants using topical or inhaled corticosteroids;
   * Short-term (≤7 days) use of glucocorticoids equivalent to ≤10 mg of prednisone daily for the prevention or treatment of non-autoimmune allergic diseases is permitted;
6. Participants with known interstitial lung disease or non-infectious pneumonia requiring systemic treatment with glucocorticoids;
7. Participants having clinically serious cardiovascular diseases (unstable angina or myocardial infarction within 6 months before enrollment), diabetes, or hypertension;
8. Participants having a history of human immunodeficiency virus infection, or having other acquired or congenital immunodeficiency diseases, or having a history of organ transplantation;
9. Patients with active chronic hepatitis B or active hepatitis C. Hepatitis B virus carriers, stable hepatitis B after drug treatment (DNA titer not higher than 500 IU/mL or copy number <1000 copies/ml) and cured hepatitis C patients (HCV RNA test negative) can be enrolled;
10. Participants having a serious infection within 4 weeks before the first administration of HX009, or having an active infection that require oral or intravenous antibiotic treatment;
11. Participants having severe allergic reactions to macromolecular protein preparations/monoclonal antibodies, or to any drug component of HX009 (CTCAE 5.0 grade greater than 3);
12. Participated in other drug clinical trials within 4 weeks before the first administration of HX009;
13. Alcohol dependent or known history of drug abuse within the past year;
14. Participants with poor compliance due to known history of neurological or mental disorders, such as epilepsy, dementia;
15. Pregnant or breastfeeding women;
16. Participants with pleural effusion, abdominal effusion or pericardial effusion with clinical symptoms;
17. Those who have received blood transfusion therapy within 4 weeks before the start of treatment or received hematopoietic stimulating factor therapy within 2 weeks, such as colony stimulating factor, erythropoietin, thrombopoietin, etc.;
18. According to the investigator's judgment, the subjects have other factors that may cause them to be forced to terminate the study halfway, such as serious diseases requiring concomitant treatment, family or social factors, which may affect the safety of the subjects or the collection of experimental data.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2021-05-12 (Actual); Primary Completion 2022-12-10 (Estimated); Study Completion 2023-02-10 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) of patients with solid tumors treated with HX009 assessed by the Independent Review Committee (IRC) | Approximately 1 year
  The ORR is defined as the percentage of participants in the analysis population who had a confirmed Complete Response or Partial Response using RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Objective response rate(ORR) of patients with solid tumors treated with HX009 per Investigator Assessment | Approximately 1 year
  The ORR is defined as the percentage of participants in the analysis population who had a confirmed Complete Response or Partial Response using RECIST 1.1 criteria.
Duration of response (DoR) of patients with solid tumors treated with HX009 | Approximately 1 year
  The DoR is defined as the time from the first recorded response (CR or PR) to the first recorded tumor progression or death due to any cause.
Disease control rate (DCR) of patients with solid tumors treated with HX009 | Approximately 1 year
  The DCR is defined as the percentage of participants in the analysis population who had a confirmed Complete Response, or Partial Response, or Stable Disease using RECIST 1.1 criteria.
Progression-free survival (PFS) of patients with solid tumors treated with HX009 | Approximately 1 year
  PFS is defined as the time from the start of the first dose and the first documented disease progression using RECIST 1.1 criteria or death of any cause.
Overall survival (OS) of patients with solid tumors treated with HX009 | Approximately 1 year
  OS is defined as the time between the start of the first dose and death of any cause.
Incidence of treatment-related adverse events in patients with advanced solid tumors treated with HX009 | AEs will be collected from the start of the study treatment up to 90 days after the last dose.
  Adverse events (AEs) related to HX009 as determined by the investigator are recorded and graded according to the Common Terminology Criteria for Adverse Events (CTCAE - Version 5.0).
Severity of treatment-related adverse events in patients with advanced solid tumors treated with HX009 | AEs will be collected from the start of the study treatment up to 90 days after the last dose.
  Adverse events (AEs) related to HX009 as determined by the investigator are recorded and graded according to the Common Terminology Criteria for Adverse Events (CTCAE - Version 5.0).
Number of patients having detectable anti-drug antibody (ADA) of HX009 | Approximately 1 year
  Detection of ADA is a measure of immunogenicity of HX009
Number of patients having detectable neutralizing antibody (Nab) of HX009 | Approximately 1 year
  Detection of Nab is a measure of immunogenicity of HX009
Elimination half-life (t1/2β) of HX009 in patients with advanced solid tumors | Approximately 1 year
  Key pharmacokinetic parameter
Mean residence time in the body (MRT) of HX009 in patients with advanced solid tumors | Approximately 1 year
  Key pharmacokinetic parameter
Area under the concentration-time curve (AUC0-t) of HX009 in patients with advanced solid tumors | Approximately 1 year
  Key pharmacokinetic parameter
Peak plasma concentration (Cmax) of HX009 in patients with advanced solid tumors | Approximately 1 year
  Key pharmacokinetic parameter
Time to peak plasma concentration (Tmax) of HX009 in patients with advanced solid tumors | Approximately 1 year
  Key pharmacokinetic parameter

CONTACTS AND LOCATIONS:
Overall Officials: Jing Huang, MD, Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Shenzhen Center, Shenzhen, Guangdong, China